CLINICAL TRIAL: NCT03804710
Title: A Clinical Study to Investigate the Effects of Two Developmental Cosmetic Moisturizing Cream Formulations on the Barrier Function of Human Skin on the Face and Legs
Brief Title: To Evaluate the Effect of Moisturizing Creams on Skin Barrier Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 209638
Record Dates: First submitted 2019-01-11; First posted 2019-01-15 (Actual); Results first posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Dry Skin; Skin Care
Keywords: Skin care, Moisturizing Cream

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test Product 1 (Experimental): Participants will apply 2 pumps of the test product (approximately 0.3ml x 2= 0.6ml) to the randomly assigned side of the face, including forehead and chin, and 6 pumps of test product (approximately 0.3 ml x 6 = 1.8 ml) to the randomly assigned lower leg (below the knee; above the ankle) topically twice-daily (in the morning and evening) after cleansing.
  Interventions: Drug: Developmental moisturizing cream 1
- Test Product 2 (Experimental): Participants will apply pea-sized amount of the test product (approximately 0.6ml) to the randomly assigned side of the face, including forehead and chin, and walnut-sized amount of the test product (approximately 1.8 ml) to the randomly assigned lower leg (below the knee; above the ankle) twice-daily (in the morning and evening) after cleansing.
  Interventions: Drug: Developmental moisturizing cream 2
- Standard soap cleanser (Placebo Comparator): Participants will use wet soap with warm water and form lather. Participants will cleanse their entire face and both lower legs (between the knees and ankles) twice daily (morning and evening).
  Interventions: Other: Standard cleanser soap

INTERVENTIONS:
Drug: Developmental moisturizing cream 1 — Participants will topically apply developmental moisturizing cream 1
  Arms: Test Product 1
Drug: Developmental moisturizing cream 2 — Participants will topically apply developmental moisturizing cream 2
  Arms: Test Product 2
Other: Standard cleanser soap — Participants will cleanse the entire face and both lower legs (between the knees and the ankles)with simple pure soap
  Arms: Standard soap cleanser

SUMMARY:
The aim of this study is to evaluate the impact of twice-daily topical application of two different moisturizing creams on skin barrier function for 4 weeks.

DETAILED DESCRIPTION:
This study will be a randomized, evaluator-blind, single-center, two-treatment regimen, controlled, parallel-group, with a treatment period of 4 weeks. The study will assess the skin barrier function of the two-treatment regimen in healthy participants with dry, sensitive skin on the face and lower legs. All participants will be centrally randomized to one of the 2 treatment groups using an Interactive Response Technology (IRT).

ELIGIBILITY:
Inclusion Criteria:

1. Participant provision of a signed and dated informed consent document indicating that the participant has been informed of all pertinent aspects of the study before any assessment is performed.
2. A participant who is willing and able to comply with scheduled visits, the product application schedule, the Lifestyle Considerations, and other study procedures which includes: a) to remove facial make-up at the screening visit to allow visual assessments; b) using other skin-care products is not permitted including but not limited to: leave-on cosmetics, moisturizers, lotions, creams, sunscreens, soaps, cleansing, exfoliation products, etc. on their face or legs, other than the standard soap and study product(s) provided; c) at all post baseline study visit days, participants must cleanse their face and legs with the standard soap and then apply the test product (s) approximately 10-16 hours before each study appointment (i.e. evening before); d) no use of any product on the face or legs, including the standard soap and test product, within 10 hours of all instrumental measurements on visit days (no showering/bathing permitted with soaps/shampoo within this period) will be permitted.
3. A participant in good general and mental health with, in the opinion of the investigator or medically qualified designee (if the investigator is not suitably qualified), no clinically significant/relevant abnormalities in medical history or upon dermatologist examination, or condition, that would impact the participant's safety, wellbeing or the outcome of the study, if they were to participate in the study, or affect the individual's ability to understand and follow study procedures and requirements.
4. A participant who responds "Yes" to the following question: Do you consider yourself to have dry, sensitive skin on your face and very dry skin on your legs?
5. A participant with an overall dryness assessment total score of ≥3 for each side of the face at screening visit (Visit 1) and baseline visit (Visit 2). With no more than 0.5-unit score difference between each side of the face. Including an examiner score of at ≥ 1 (slight) for the roughness parameter.
6. A participant with an overall dryness assessment total score of ≥6 for each leg at screening visit (Visit 1) and baseline visit (Visit 2). With no more than 1-unit score difference between each leg.
7. A participant with a Fitzpatrick skin type I-IV.

Exclusion Criteria:

1. A participant who is an employee of the investigational site, either directly involved in the conduct of the study or a member of their family; or an employee of the investigational site otherwise supervised by the investigator; or, a GSK CH employee directly involved in the conduct of the study or a member of their immediate family.
2. A participant who has participated in other studies (including non-medicinal studies) involving investigational product(s) within 30 days prior to study entry and/or during study participation.
3. A participant with, in the opinion of the investigator or medically qualified designee, an acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product application or may interfere with the interpretation of study results and, in the judgment of the investigator or medically qualified designee, would make the participant inappropriate for entry into this study.
4. A female participant who is pregnant (self-reported) or intending to become pregnant.
5. A female participant who is breastfeeding.
6. A participant with known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
7. A participant who, in the opinion of the investigator or medically qualified designee, should not participate in the study.
8. A participant with current or recent (within 6 months before the start of the study) history of atopic lesions and/or eczema.
9. A participant with a history of allergic reactions to topical-use products, cosmetics or medications or their ingredients.
10. A participant with any history of significant diseases or medical conditions known to alter skin or eye appearance or physiologic response (e.g. Type 2 diabetes) which could, in the opinion of the Investigator, preclude topical application of the investigational products and/or interfere with the evaluation of the test site reaction.
11. A participant presenting open sores, pimples, or cysts at the application site (face or lower legs).
12. A participant with an active dermatosis (local or disseminated) that might interfere with the results of the study.
13. A participant currently using any medication which in the opinion of the investigator, may affect the evaluation of the investigational product, or place the participant at undue risk
14. A participant who has used any of the following topical or systemic medications up to 1 month before the screening visit or intends to use during the study period: immuno-suppressants, antihistamines, non-steroidal anti-inflammatory drugs (NSAIDS), and corticosteroids.
15. A participant who has used oral or topical treatment with vitamin A acid and/or its derivatives up to 1 month before the screening visit or intends to use during the study period.
16. A participant who intends to use any topical drug or medication on the proposed application areas. A participant who has been vaccinated up to 1 month before the screening visit or is intending to receive a vaccination during their participation in the study.

18. A participant currently receiving allergy injections, or received an allergy injection within 7 days prior to Visit 1, or expects to begin injections during study participation 19. A participant with a recent history (within the last 5 years) of alcohol or other substance abuse.

20. A participant with any skin marks on the face or lower legs that might interfere with the evaluation of possible skin reactions (e.g. pigmentation disorders, vascular malformations, scars, tattoos, excessive hair, numerous freckles). 21. Participants with corneal ulcers, keratoconus, blepharitis, meibomitis, pterygium, chemosis, moderately or severe hyperemia or other active ocular diseases. 22. A participant who has previously been enrolled in this study. 23. A participant who is unwilling to abstain from smoking tobacco or using any other nicotine containing products.

24. A participant with visible sunburn on any of the test sites. 25. A participant with moles, tattoos, scars, hairs, etc. at the test areas if it is likely that they could affect the assessments. 26. A participant who has used self-tanning products on the test areas (face and arms) within 2 weeks prior to the screening visit. 27. A participant who intends to expose their skin to natural or artificial ultraviolet (UV) light (e.g.

sunbathing or tanning beds). 28. A participant with any participant self-assessed or dermatologist dryness parameter score 4 (very severe) on the test areas of the lower legs or face.

29. Any participant who, in the judgment of the Investigator, should not participate in the study.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 158 (Actual)
Dates: Start 2019-01-22 (Actual); Primary Completion 2019-04-16 (Actual); Study Completion 2019-04-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline (for GlaxoSmithKline; Human Genome Sciences Inc., a GSK Company; Sirtris, a GSK Company; Stiefel, a GSK Company; ViiV Healthcare)
Locations (1):
- GSK Investigational Site, Schenefeld, Schleswig-Holstein, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were enrolled at one center in Germany.
Pre-assignment Details: A total 174 participants were screened, out of which 158 participants were enrolled, 149 participants were randomized and 25 participants not randomized. Out of 149 randomized participants, 7 participants did not completed study because 3 participants experienced adverse event, 3 participants withdrew consent and 1 participant due to other reason.
Groups:
- Treatment Regimen 1 (Test Product 1 + Standard Soap): Participants randomized to this treatment regimen and were further randomized within regimen left and right side in equal proportion. Participants applied allocated test product 1 topically, (approximately 0.3 milliliter (mL) × 2 pumps = 0.6 mL, each pump contains 0.3 mL) on face and (approximately 0.3 mL × 6 pumps = 1.8 mL, each pump contains 0.3 mL) on leg after cleansing with standard cleanser (simple pure soap), to the designated side per randomization, the same side of the face including forehead and chin and the same leg (left or right), twice a day (morning and evening) for 4 weeks. Morning and evening applications were separated by approximately 8 to 12 hours (hrs).
- Treatment Regimen 2 (Test Product 2 + Standard Soap): Participants randomized to this treatment regimen and were further randomized within regimen left and right side in equal proportion. Participants applied allocated test product 2 topically, (approximately 0.3 mL × 2 pumps = 0.6 mL, each pump contains 0.3 mL) on face and (approximately 0.3 mL × 6 pumps = 1.8 mL, each pump contains 0.3 mL) on leg after cleansing with standard cleanser (simple pure soap), to the designated side per randomization, the same side of the face including forehead and chin and the same leg (left or right), twice a day (morning and evening) for 4 weeks. Morning and evening applications were separated by approximately 8 to 12 hrs.
Period: Overall Study
Arm/Group | Treatment Regimen 1 (Test Product 1 + Standard Soap) | Treatment Regimen 2 (Test Product 2 + Standard Soap)
Started | 75 | 74
Completed | 73 | 69
Not Completed | 2 | 5
Not completed — Adverse Event | 0 | 3
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population comprised of all randomized participants who applied at least one dose of the study product.
Groups:
- Treatment Regimen 1 (Test Product 1 + Standard Soap): Participants randomized to this treatment regimen and were further randomized within regimen left and right side in equal proportion. Participants applied allocated test product 1 topically, (approximately 0.3 mL × 2 pumps = 0.6 mL, each pump contains 0.3 mL) on face and (approximately 0.3 mL × 6 pumps = 1.8 mL, each pump contains 0.3 mL) on leg after cleansing with standard cleanser (simple pure soap), to the designated side per randomization, the same side of the face including forehead and chin and the same leg (left or right), twice a day (morning and evening) for 4 weeks. Morning and evening applications were separated by approximately 8 to 12 hrs.
- Treatment Regimen 2 (Test Product 2 + Standard Soap): Participants randomized to this treatment regimen and were further randomized within regimen left and right side in equal proportion. Participants randomized to this treatment regimen and were further randomized within regimen left and right side. Participants applied allocated test product 2 topically, (approximately 0.3 mL × 2 pumps = 0.6 mL, each pump contains 0.3 mL) on face and (approximately 0.3 mL × 6 pumps = 1.8 mL, each pump contains 0.3 mL) on leg after cleansing with standard cleanser (simple pure soap), to the designated side per randomization, the same side of the face including forehead and chin and the same leg (left or right), twice a day (morning and evening) for 4 weeks. Morning and evening applications were separated by approximately 8 to 12 hrs.
- Total: Total of all reporting groups
Arm/Group | Treatment Regimen 1 (Test Product 1 + Standard Soap) | Treatment Regimen 2 (Test Product 2 + Standard Soap) | Total
Number analyzed (Participants) | 75 | 74 | 149
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.8 (9.64) | 49.6 (11.98) | 51.2 (10.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 74 | 149
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/African Heritage | 0 | 0 | 0
  American Indian or Alaskan Native | 0 | 0 | 0
  Asian - Central/South Asian Heritage | 1 | 0 | 1
  Asian - East Asian Heritage | 0 | 0 | 0
  Asian - Japanese Heritage | 0 | 0 | 0
  Asian - South East Asian Heritage | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  White - Arabic/North African Heritage | 1 | 1 | 2
  White - White/Caucasian/European Heritage | 73 | 73 | 146
Fitzpatrick Skin Type Grading [Count of Participants; unit: Participants] — Fitzpatrick scale was used to classify a participant's skin type by their response to sun exposure. This scale emphasizes on potentials for irritation, burns and hyperpigmentation, indicators for future product choices. This scale has six grading, where I refers to always burns easily; never tans, II refers to always burns easily; tans minimally, III refers to burns moderately; tans gradually, IV refers to burns minimally, always tans well, V refers to rarely burns, tans profusely and VI refers to never burns.
  Participants
    I - Pale white skin | 5 | 4 | 9
    II - White skin | 35 | 32 | 67
    III - Light brown skin | 33 | 35 | 68
    IV - Moderate brown skin | 2 | 3 | 5
    V - Dark brown skin | 0 | 0 | 0
    VI - Deeply pigmented dark brown to black skin | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Trans-epidermal Water Loss (TEWL) Following Application of Test Regimen on Face (Area 1 Compared to Area 2) at Day 29
Description: TEWL was measured using the Tewameter TM 300. TEWL is a non-invasive method to measure the integrity of stratum corneum barrier function. Tewameter probe measures the density gradient of the water evaporation from the skin indirectly by two pairs of sensors (temperature and relative humidity) inside a hollow cylinder. The probe was held in place on the skin for one measurement, for 40 sec, to ensure that a stable value has been established. The values of the last 10 sec are averaged as the actual measurement values. An increase in TEWL values shows damage to the skin barrier function. TEWL was measured at area 1 (right face) and 2 (left face) at baseline visit (Visit 2) prior to any study product application and then measured throughout the study period per the study schedule. Change from baseline was calculated as the value at specified visit (Visit 5/Day 29) minus the baseline value.
Time Frame: Baseline and Day 29
Population: Modified Intent-to-Treat (MITT) population. Here, number analyzed indicates participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: g/m^2/hr
Groups:
- Test Product 1: Participants randomized to this treatment regimen and were further randomized within regimen left and right side in equal proportion. Participants applied allocated test product 1 topically, (approximately 0.3 ml x 2 pumps = 0.6 ml, each pump contains 0.3 ml) on face and (approximately 0.3 ml x 6 pumps = 1.8 ml, each pump contains 0.3 ml) on leg after cleansing with standard cleanser to designated side per randomization, the same side of face including forehead and chin and the same leg (left or right), twice a day (morning and evening) for 4 weeks. Morning and evening applications were separated by approximately 8 to 12 hrs.
- Test Product 2: Participants randomized to this treatment regimen and were further randomized within regimen left and right side in equal proportion. Participants applied allocated test product 2 topically, (approximately 0.3 ml x 2 pumps = 0.6 ml, each pump contains 0.3 ml) on face and (approximately 0.3 ml x 6 pumps = 1.8 ml, each pump contains 0.3 ml) on leg after cleansing with standard cleanser to designated side per randomization, the same side of face including forehead and chin and the same leg (left or right), twice a day (morning and evening) for 4 weeks. Morning and evening applications were separated by approximately 8 to 12 hrs.
- Standard Cleanser Soap: Standard cleanser (Simple pure soap) utilized for cleansing face and leg before application of either test product 1 or product 2 topically, twice a day (morning and evening) for 4 weeks. Morning and evening applications were separated by approximately 8 to 12 hrs.
Arm/Group | Test Product 1 | Test Product 2 | Standard Cleanser Soap
Number analyzed (Participants) | 70 | 66 | 137
g/m^2/hr | -5.077 (6.4082) | -4.946 (6.2628) | -3.692 (6.0635)

2. Secondary Outcome: Change From Baseline in TEWL Following Application of Test Regimen on Legs (Area 5 Compared to Area 6) at Day 29
Description: TEWL was measured using the Tewameter TM 300. TEWL is a non-invasive method to measure the integrity of stratum corneum barrier function. Tewameter probe measures the density gradient of the water evaporation from the skin indirectly by two pairs of sensors (temperature and relative humidity) inside a hollow cylinder. The probe was held in place on the skin for one measurement, for 40 sec, to ensure that a stable value has been established. The values of the last 10 sec are averaged as the actual measurement values. An increase in TEWL values shows damage to the skin barrier function. TEWL was measured at area 5 (right leg) and 6 (left leg) at baseline visit (Visit 2) prior to any study product application and then measured throughout the study period per the study schedule. Change from baseline was calculated as the value at specified visit (Visit 5/Day 29) minus the baseline value (Visit 2).
Time Frame: Baseline and Day 29
Population: MITT Population. Here, number analyzed indicates participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: g/m^2/hr
Arm/Group | Test Product 1 | Test Product 2 | Standard Cleanser Soap
Number analyzed (Participants) | 71 | 66 | 137
g/m^2/hr | -3.582 (3.7399) | -3.153 (3.0987) | -1.321 (4.0207)

3. Secondary Outcome: Change From Baseline in TEWL Following Application of Test Regimen on Face (Area 1 Compared to Area 2) at Day 15
Description: TEWL was measured using the Tewameter TM 300. TEWL is a non-invasive method to measure the integrity of stratum corneum barrier function. Tewameter probe measures the density gradient of the water evaporation from the skin indirectly by two pairs of sensors (temperature and relative humidity) inside a hollow cylinder. The probe was held in place on the skin for one measurement, for 40 sec, to ensure that a stable value has been established. The values of the last 10 sec are averaged as the actual measurement values. An increase in TEWL values shows damage to the skin barrier function. TEWL was measured at area 1 (right face) and 2 (left face) at baseline visit (Visit 2) prior to any study product application and then measured throughout the study period per the study schedule. Change from baseline was calculated as the value at specified visit (Visit 5/Day 29) minus the baseline value (Visit 2).
Time Frame: Baseline and Day 15
Population: MITT Population. Here, number analyzed indicates participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: g/m^2/hr
Arm/Group | Test Product 1 | Test Product 2 | Standard Cleanser Soap
Number analyzed (Participants) | 72 | 68 | 140
g/m^2/hr | -4.474 (6.2645) | -5.963 (7.0847) | -3.297 (5.5348)

4. Secondary Outcome: Change From Baseline in TEWL Following Application of Test Regimen on Legs (Area 5 Compared to Area 6) at Day 15
Description: as for outcome 2
Time Frame: Baseline and Day 15
Population: MITT Population. Here, number analyzed indicates participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: g/m^2/hr
Arm/Group | Test Product 1 | Test Product 2 | Standard Cleanser Soap
Number analyzed (Participants) | 72 | 68 | 140
g/m^2/hr | -2.070 (3.0035) | -1.944 (3.3337) | -0.708 (3.2338)

5. Secondary Outcome: Change From Baseline in Corneometer Values Following Application of Test Regimen on Face (Area 1 Compared to Area 2) at Two Different Time-points [30 Minutes (Mins) and 6 Hrs After First Application] at Day 1 and One Time-point at Day 2
Description: Stratum corneum (SC) moisturization measured using the Corneometer CM 825. The measuring principle is based on changes in the capacitance of the measuring head, functioning as condensator. The electric field was created between gold conductors to enable the dielectricity of the SC to be measured. Because the dielectricity varies as a function of the skin's water content, the SC moisturization was measured. Corneometer probe was placed in contact with the skin of the participants test site for 1 to 2 sec per measurement. The measurement will be taken 5 times in total and then an average reading will be calculated for each site and time point. The Corneometer values lower than 30 international units (i.u) represent very dry skin and values between 30 to 50 i.u represent dry skin on the forearm. Higher value of Corneometer indicates high moisture content. The area 1 (right face) and area 2 (left face) were considered.
Time Frame: Baseline, 30 mins and 6 hrs after first treatment application on Day 1 and 24 hrs after treatment application on Day 2
Population: MITT Population. Here, number analyzed indicates participants with available data for this outcome measure. Baseline value is the value obtained on Day 1 (Visit 2) before study product application for Corneometer variable. Change from Baseline was calculated as the value at specified visit minus the Baseline value.
Measure: Mean (Standard Deviation); unit: International units (i.u.)
Arm/Group | Test Product 1 | Test Product 2 | Standard Cleanser Soap
Number analyzed (Participants) | 75 | 74 | 149
International units (i.u.)
  Day 1, 30 mins, post-dose | 24.628 (8.8144) | 12.048 (9.3662) | 0.246 (5.4461)
  Day 1, 6 hrs | 14.756 (8.3951) | 6.760 (7.3969) | -0.381 (6.8182)
  Day 2, Visit 3: number analyzed (Participants) | 73 | 74 | 147
  Day 2, Visit 3 | 3.032 (7.5869) | 1.707 (6.5054) | -1.765 (7.7254)

6. Secondary Outcome: Change From Baseline in Corneometer Values Following Application of Test Regimen on Legs (Area 5 Compared to Area 6) at Two Different Time-points (30 Mins and 6 Hrs After First Application) at Day 1 and One Time-point at Day 2
Description: SC moisturization measured using the Corneometer CM 825. The measuring principle is based on changes in the capacitance of the measuring head, functioning as condensator. The electric field was created between gold conductors to enable the dielectricity of the SC to be measured. Because the dielectricity varies as a function of the skin's water content, the SC moisturization was measured. Corneometer probe was placed in contact with the skin of the participants test site for 1 to 2 sec per measurement. The measurement will be taken 5 times in total and then an average reading will be calculated for each site and time point. The Corneometer values lower than 30 i.u represent very dry skin and values between 30 to 50 i.u represent dry skin on the forearm. Higher value of Corneometer indicates high moisture content. The area 5 (right leg) and area 6 (left leg) were considered.
Time Frame: Baseline, Day 1 and Day 2
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: i.u.
Arm/Group | Test Product 1 | Test Product 2 | Standard Cleanser Soap
Number analyzed (Participants) | 75 | 74 | 149
i.u.
  Day 1, 30 mins, post-dose | 9.636 (5.6719) | 7.537 (5.1710) | -0.934 (2.5630)
  Day 1, 6 hrs | 0.762 (5.2888) | 0.096 (5.0023) | -7.120 (3.6854)
  Day 2, Visit 3: number analyzed (Participants) | 73 | 74 | 147
  Day 2, Visit 3 | 2.116 (5.1318) | 0.685 (5.2522) | -2.341 (4.8045)

7. Secondary Outcome: Change From Baseline in Corneometer Values Following Application of Test Regimen on Face (Area 1 Compared to Area 2) at Day 15 and 29
Description: SC moisturization measured using the Corneometer CM 825. The measuring principle is based on changes in the capacitance of the measuring head, functioning as condensator. The electric field was created between gold conductors to enable the dielectricity of the SC to be measured. Because the dielectricity varies as a function of the skin's water content, the SC moisturization was measured. Corneometer probe was placed in contact with the skin of the participants test site for 1 to 2 sec per measurement. The measurement will be taken 5 times in total and then an average reading will be calculated for each site and time point. The Corneometer values lower than 30 i.u represent very dry skin and values between 30 to 50 i.u represent dry skin on the forearm. Higher value of Corneometer indicates high moisture content. The area 1 (right face) and area 2 (left face) were considered.
Time Frame: Baseline, Day 15 and 29
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: i.u.
Arm/Group | Test Product 1 | Test Product 2 | Standard Cleanser Soap
Number analyzed (Participants) | 75 | 74 | 149
i.u.
  Day 15, Visit 4: number analyzed (Participants) | 72 | 68 | 140
  Day 15, Visit 4 | 11.448 (9.6078) | 11.517 (8.4413) | 1.454 (8.5126)
  Day 29, Visit 5: number analyzed (Participants) | 70 | 66 | 137
  Day 29, Visit 5 | 13.573 (9.6777) | 11.870 (7.8857) | 3.506 (8.4246)

8. Secondary Outcome: Change From Baseline in Corneometer Values Following Application of Test Regimen on Legs (Area 5 Compared to Area 6) at Day 15 and 29
Description: as for outcome 6
Time Frame: Baseline, Day 15 and Day 29
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: i.u.
Arm/Group | Test Product 1 | Test Product 2 | Standard Cleanser Soap
Number analyzed (Participants) | 75 | 74 | 149
i.u.
  Day 15, Visit 4: number analyzed (Participants) | 72 | 68 | 140
  Day 15, Visit 4 | 8.538 (6.3133) | 7.452 (6.7550) | -1.094 (5.9129)
  Day 29, Visit 5: number analyzed (Participants) | 71 | 66 | 137
  Day 29, Visit 5 | 8.443 (7.6121) | 8.944 (8.5479) | -1.273 (6.7258)

9. Secondary Outcome: Change From Baseline in TEWL Following Application of Test Regimen on Face (Area 1 Compared to Area 2) at Day 30, 31, 32, 33 and 34
Description: as for outcome 1
Time Frame: Baseline, Day 30, 31, 32, 33 and 34
Population: MITT Population. Here, number analyzed indicates participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: g/m^2/hr
Arm/Group | Test Product 1 | Test Product 2 | Standard Cleanser Soap
Number analyzed (Participants) | 75 | 74 | 149
g/m^2/hr
  Day 30, Visit 6: number analyzed (Participants) | 71 | 69 | 141
  Day 30, Visit 6 | -4.556 (6.4520) | -3.998 (6.3336) | -3.045 (6.3823)
  Day 31, Visit 7: number analyzed (Participants) | 70 | 69 | 140
  Day 31, Visit 7 | -3.521 (7.0138) | -4.100 (6.3224) | -2.884 (6.2981)
  Day 32, Visit 8: number analyzed (Participants) | 71 | 68 | 140
  Day 32, Visit 8 | -3.280 (6.8111) | -3.219 (7.3358) | -2.293 (6.2826)
  Day 33, Visit 9: number analyzed (Participants) | 71 | 69 | 141
  Day 33, Visit 9 | -2.127 (7.5335) | -3.538 (6.4934) | -2.401 (6.5692)
  Day 34, Visit 10: number analyzed (Participants) | 71 | 69 | 141
  Day 34, Visit 10 | -2.292 (7.1913) | -3.270 (6.8906) | -2.572 (6.9373)

10. Secondary Outcome: Change From Baseline in TEWL Following Application of Test Regimen on Legs (Area 5 Compared to Area 6) at Day 30, 31, 32, 33 and 34
Description: TEWL was measured using the Tewameter TM 300. TEWL is a non-invasive method to measure the integrity of stratum corneum barrier function. Tewameter probe measures the density gradient of the water evaporation from the skin indirectly by two pairs of sensors (temperature and relative humidity) inside a hollow cylinder. The probe was held in place on the skin for one measurement, for 40 sec, to ensure that a stable value has been established. The values of the last 10 sec are averaged as the actual measurement values. An increase in TEWL values shows damage to the skin barrier function. TEWL was measured at area 5 (right leg) and 6 (left leg) at baseline visit (Visit 2) prior to any study product application and then measured throughout the study period per the study schedule. Change from baseline was calculated as the value at specified visit (Visit 5/Day 29) minus the baseline value.
Time Frame: Baseline, Day 30, 31, 32, 33 and 34
Population: MITT Population. Here, number analyzed indicates participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: g/m^2/hr
Arm/Group | Test Product 1 | Test Product 2 | Standard Cleanser Soap
Number analyzed (Participants) | 75 | 74 | 149
g/m^2/hr
  Day 30, Visit 6: number analyzed (Participants) | 73 | 69 | 142
  Day 30, Visit 6 | -3.521 (4.7730) | -3.061 (3.0287) | -1.400 (4.3060)
  Day 31, Visit 7: number analyzed (Participants) | 72 | 69 | 141
  Day 31, Visit 7 | -3.466 (5.5323) | -2.752 (5.0402) | -1.399 (4.1302)
  Day 32, Visit 8: number analyzed (Participants) | 73 | 68 | 141
  Day 32, Visit 8 | -3.873 (3.7703) | -3.237 (3.6959) | -1.320 (3.7519)
  Day 33, Visit 9: number analyzed (Participants) | 73 | 69 | 142
  Day 33, Visit 9 | -3.293 (5.9573) | -3.348 (3.3339) | -0.813 (4.5829)
  Day 34, Visit 10: number analyzed (Participants) | 73 | 69 | 142
  Day 34, Visit 10 | -3.474 (5.2560) | -3.327 (3.4768) | -0.991 (3.7641)

11. Secondary Outcome: Change From Baseline in Corneometer Values Following Application of Test Regimen on Face (Area 1 Compared to Area 2) at Day 30, 31, 32, 33 and 34
Description: as for outcome 7
Time Frame: Baseline, Day 30, 31, 32, 33 and 34
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: i.u.
Arm/Group | Test Product 1 | Test Product 2 | Standard Cleanser Soap
Number analyzed (Participants) | 75 | 74 | 149
i.u.
  Day 30, Visit 6: number analyzed (Participants) | 71 | 69 | 141
  Day 30, Visit 6 | 7.279 (8.0036) | 7.175 (8.4301) | 2.927 (8.0479)
  Day 31, Visit 7: number analyzed (Participants) | 70 | 69 | 140
  Day 31, Visit 7 | 5.581 (7.6171) | 4.441 (8.3006) | 1.866 (8.1570)
  Day 32, Change at visit 8: number analyzed (Participants) | 71 | 68 | 140
  Day 32, Change at visit 8 | 3.948 (8.6287) | 1.823 (8.0040) | 0.829 (8.7018)
  Day 33, Visit 9: number analyzed (Participants) | 71 | 69 | 141
  Day 33, Visit 9 | 2.839 (9.0299) | 1.772 (7.9661) | 0.608 (9.6741)
  Day 34, Visit 10: number analyzed (Participants) | 71 | 69 | 141
  Day 34, Visit 10 | 1.965 (10.0299) | 1.686 (7.5388) | 0.682 (9.2882)

12. Secondary Outcome: Change From Baseline in Corneometer Values Following Application of Test Regimen on Legs (Area 5 Compared to Area 6) at Day 30, 31, 32, 33 and 34
Description: as for outcome 6
Time Frame: Baseline, Day 30, 31, 32, 33 and 34
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: i.u.
Arm/Group | Test Product 1 | Test Product 2 | Standard Cleanser Soap
Number analyzed (Participants) | 75 | 74 | 149
i.u.
  Day 30, Visit 6: number analyzed (Participants) | 73 | 69 | 142
  Day 30, Visit 6 | 4.738 (6.9914) | 5.372 (7.1154) | -2.692 (6.6993)
  Day 31, Visit 7: number analyzed (Participants) | 72 | 69 | 141
  Day 31, Visit 7 | 2.943 (6.6218) | 5.843 (7.3787) | -2.223 (6.9870)
  Day 32, Visit 8: number analyzed (Participants) | 73 | 68 | 141
  Day 32, Visit 8 | 2.549 (6.8103) | 4.054 (6.8908) | -2.673 (6.4090)
  Day 33, Visit 9: number analyzed (Participants) | 73 | 69 | 142
  Day 33, Visit 9 | 2.135 (6.1634) | 3.939 (7.9278) | -2.732 (6.0150)
  Day 34, Visit 10: number analyzed (Participants) | 73 | 74 | 142
  Day 34, Visit 10 | 3.894 (6.3960) | 5.627 (7.2834) | -0.942 (6.8374)

13. Secondary Outcome: Change From Pre-challenge in TEWL Following Application of Test Regimen on Face (Area 3 Compared to Area 4) at 3 Different Time Points of Strips Removal (3,6 and 9) at Day 29
Description: Tape-stripping method was used to evaluate the impact of physical challenge to the skin barrier after product use. Stripping challenge was performed on D-Squame sites on area 3 (right face) and area 4 (left face) at Day 29 by sequential application and removal of D-Squame adhesive 3, 6, and 9 discs. A Series of D-Squame discs were applied over the areas with uniform pressure for 5 sec with a stamp to ensure consistent adhesion to the skin. The disc was pulled off the skin with one fluent and decisive movement. TEWL was measured pre-challenge and after 3, 6, and 9 discs had been removed. TEWL was measured using the Tewameter TM 300. Tewameter probe measures the density gradient of the water evaporation from the skin indirectly by two pairs of sensors (temperature and relative humidity) inside a hollow cylinder. TEWL measurement was taken in triplicate. The average reading was considered for each area and time point. An increase in TEWL values shows damage to the skin barrier function.
Time Frame: Day 31
Population: MITT Population. Here, number analyzed indicates participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: g/m^2/hr
Arm/Group | Test Product 1 | Test Product 2 | Standard Cleanser Soap
Number analyzed (Participants) | 75 | 74 | 149
g/m^2/hr
  Removal of 3 tape strips: number analyzed (Participants) | 70 | 66 | 137
  Removal of 3 tape strips | 5.52 (5.762) | 4.86 (3.339) | 5.59 (4.421)
  Removal of 6 tape strips: number analyzed (Participants) | 70 | 66 | 137
  Removal of 6 tape strips | 15.64 (11.883) | 14.28 (10.510) | 17.46 (11.698)
  Removal of 9 tape strips: number analyzed (Participants) | 70 | 66 | 137
  Removal of 9 tape strips | 27.18 (16.425) | 24.33 (14.524) | 30.74 (16.715)

14. Secondary Outcome: Change From Pre-challenge in TEWL Following Application of Test Regimen on Legs (Area 7 Compared to Area 8) at 3 Different Time Points of Strips Removal (4, 8 and 12) at Day 29
Description: Tape-stripping method was used to evaluate the impact of a physical challenge to the skin barrier after product use. Stripping challenge was performed on D-Squame sites on area 3 (right face) and area 4 (left face) at Day 29 by sequential application and removal of D-Squame adhesive 3, 6, and 9 discs. A Series of D-Squame discs were applied over the areas with uniform pressure for 5 sec with a stamp to ensure consistent adhesion to the skin. The disc was pulled off the skin with one fluent and decisive movement. TEWL was measured pre-challenge after 3, 6, and 9 discs have been removed. TEWL was measured using the Tewameter TM 300. Tewameter probe measures the density gradient of the water evaporation from the skin indirectly by two pairs of sensors (temperature and relative humidity) inside a hollow cylinder. TEWL measurement was taken in triplicate. The average reading was considered for each area and time point. An increase in TEWL values shows damage to the skin barrier function.
Time Frame: Pre-challenge and Day 29
Population: MITT Population. Here, number analyzed indicates participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: g/m^2/hr
Arm/Group | Test Product 1 | Test Product 2 | Standard Cleanser Soap
Number analyzed (Participants) | 71 | 66 | 149
g/m^2/hr
  Removal of 4 tape strips: number analyzed (Participants) | 71 | 66 | 137
  Removal of 4 tape strips | 0.822 (0.8750) | 0.592 (1.0522) | 1.269 (1.3704)
  Removal of 8 tape strips: number analyzed (Participants) | 71 | 66 | 137
  Removal of 8 tape strips | 2.314 (2.6847) | 1.832 (1.5725) | 3.464 (1.9604)
  Removal of 12 tape strips: number analyzed (Participants) | 71 | 66 | 137
  Removal of 12 tape strips | 3.619 (1.8322) | 3.823 (2.5310) | 6.740 (4.3941)

15. Secondary Outcome: Total Protein Content Extracted From D-Squame Discs From a Total of 9 Adhesive Discs on Face (Area 3 Compared to Area 4) at Day 29
Description: Total protein content was measured using the SquameScan 850. SquameScan 850 is an instrument used to measure the protein content extracted from the skin by D-Squame tape strips. The determination is carried out by measuring the optical absorption of the strip at 850 nanometers (nm). Value displayed in percentage (%) was proportionally related to protein content. An 18 D-Squame discs were taken from participant (two sets of 9 discs from each side of the face). The protein content was analyzed for each of the discs obtained from the D-Squame stripping on area 3 (right face) and area 4 (left face) on Day 29.
Time Frame: Day 29
Population: MITT Population.
Measure: Mean (Standard Deviation); unit: Percentage (%)
Arm/Group | Test Product 1 | Test Product 2 | Standard Cleanser Soap
Number analyzed (Participants) | 70 | 66 | 149
Percentage (%) | 91.65 (19.498) | 97.53 (20.882) | 115.36 (26.320)

16. Secondary Outcome: Total Protein Content Extracted From D-Squame Discs From a Total of 12 Adhesive Discs on Leg (Area 7 Compared to Area 8) at Day 29
Description: Total protein content was measured using the SquameScan 850. SquameScan 850 is an instrument used to measure the protein content extracted from the skin by D-Squame tape strips. The determination is carried out by measuring the optical absorption of the strip at 850 nm. Value displayed in percentage (%) was proportionally related to protein content. An 24 D-Squame discs were taken from participant (two sets of 12 discs from the two separate sites of each lower leg). The protein content was analyzed for each of the discs obtained from the D-Squame stripping on area 7 (right leg) and area 8 (left leg) on Day 29.
Time Frame: Day 29
Population: MITT Population.
Measure: Mean (Standard Deviation); unit: Percentage (%)
Arm/Group | Test Product 1 | Test Product 2 | Standard Cleanser Soap
Number analyzed (Participants) | 71 | 66 | 149
Percentage (%) | 187.33 (30.773) | 201.82 (45.288) | 228.68 (36.005)

ADVERSE EVENTS:
Time Frame: Up to Day 34
Description: Adverse event (AE) reporting was performed on the safety population (N=149). Safety population included all randomized participants who applied at least one dose of the study product. Treatment-emergent adverse events were reported as per Treatment Regimen; Treatment Regimen 1 and Treatment Regimen 2 whereas Treatment related treatment emergent adverse events were reported as per Intervention; Test Product 1, Test Product 2 and Standard Soap. All adverse events were collected and reported.
Groups:
- Treatment Regimen 1 (Test Product 1 + Standard Soap): Participants randomized to this treatment regimen and were further randomized within regimen left and right side in equal proportion. Participants applied allocated test product 1 topically, (approximately 0.3 ml x 2 pumps = 0.6 ml, each pump contains 0.3 ml) on face and (approximately 0.3 ml x 6 pumps = 1.8 ml, each pump contains 0.3 ml) on leg after cleansing with standard cleanser to designated side per randomization, the same side of face including forehead and chin and the same leg (left or right), twice a day (morning and evening) for 4 weeks. Morning and evening applications were separated by approximately 8 to 12 hrs.
- Treatment Regimen 2 (Test Product 2 + Standard Soap): Participants randomized to this treatment regimen and were further randomized within regimen left and right side in equal proportion. Participants applied allocated test product 2 topically, (approximately 0.3 ml x 2 pumps = 0.6 ml, each pump contains 0.3 ml) on face and (approximately 0.3 ml x 6 pumps = 1.8 ml, each pump contains 0.3 ml) on leg after cleansing with standard cleanser to designated side per randomization, the same side of face including forehead and chin and the same leg (left or right), twice a day (morning and evening) for 4 weeks. Morning and evening applications were separated by approximately 8 to 12 hrs.
- Test Product 1: Participants applied allocated test product 1 topically, (approximately 0.3 ml x 2 pumps = 0.6 ml, each pump contains 0.3 ml) on face and (approximately 0.3 ml x 6 pumps = 1.8 ml, each pump contains 0.3 ml) on leg to designated side per randomization, the same side of face including forehead and chin and the same leg (left or right), twice a day (morning and evening) for 4 weeks. Morning and evening applications were separated by approximately 8 to 12 hrs
- Test Product 2: Participants applied allocated test product 2 topically, (approximately 0.3 ml x 2 pumps = 0.6 ml, each pump contains 0.3 ml) on face and (approximately 0.3 ml x 6 pumps = 1.8 ml, each pump contains 0.3 ml) on leg to designated side per randomization, the same side of face including forehead and chin and the same leg (left or right), twice a day (morning and evening) for 4 weeks. Morning and evening applications were separated by approximately 8 to 12 hrs.
- Standard Soap: Participants applied standard cleanser soap (for cleansing purpose) topically before applying allocated either Test Product 1 or Test Product 2 to designated side per randomization, the same side of face including forehead and chin and the same leg (left or right), twice a day (morning and evening) for 4 weeks. Morning and evening applications were separated by approximately 8 to 12 hrs.
Arm/Group | Treatment Regimen 1 (Test Product 1 + Standard Soap) | Treatment Regimen 2 (Test Product 2 + Standard Soap) | Test Product 1 | Test Product 2 | Standard Soap
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/74 | 0/75 | 0/74 | 0/149
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/74 | 0/75 | 0/74 | 0/149
Other Adverse Events (participants affected / at risk) | 19/75 | 23/74 | 5/75 | 4/74 | 7/149
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Treatment Regimen 1 (Test Product 1 + Standard Soap) (N=75) | Treatment Regimen 2 (Test Product 2 + Standard Soap) (N=74) | Test Product 1 (N=75) | Test Product 2 (N=74) | Standard Soap (N=149)
Skin irritation (Skin and subcutaneous tissue disorders) | 2 (3) | 4 (7) | 2 (2) | 2 (2) | 4 (4) — All Treatment Emergent Adverse Events were reported by treatment regimen and only Treatment Related Treatment Emergent Adverse Events were reported per-intervention since Treatment Emergent Adverse Events were not analysed per intervention.
Rash papular (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0) | 2 (2) | 0 (0) | 1 (1) — All Treatment Emergent Adverse Events were reported by treatment regimen and only Treatment Related Treatment Emergent Adverse Events were reported per-intervention since Treatment Emergent Adverse Events were not analysed per intervention.
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1) — All Treatment Emergent Adverse Events were reported by treatment regimen and only Treatment Related Treatment Emergent Adverse Events were reported per-intervention since Treatment Emergent Adverse Events were not analysed per intervention.
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) — All Treatment Emergent Adverse Events were reported by treatment regimen and only Treatment Related Treatment Emergent Adverse Events were reported per-intervention since Treatment Emergent Adverse Events were not analysed per intervention.
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) — All Treatment Emergent Adverse Events were reported by treatment regimen and only Treatment Related Treatment Emergent Adverse Events were reported per-intervention since Treatment Emergent Adverse Events were not analysed per intervention.
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) — All Treatment Emergent Adverse Events were reported by treatment regimen and only Treatment Related Treatment Emergent Adverse Events were reported per-intervention since Treatment Emergent Adverse Events were not analysed per intervention.
Nasopharyngitis (Infections and infestations) | 4 (4) | 6 (6) | 0/0 (0) | 0/0 (0) | 0/0 (0) — All Treatment Emergent Adverse Events were reported by treatment regimen and only were not analyzed per intervention.
Oral herpes (Infections and infestations) | 0 (0) | 2 (2) | 0/0 (0) | 0/0 (0) | 0/0 (0) — All Treatment Emergent Adverse Events were reported by treatment regimen and only were not analyzed per intervention.
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0) | 0/0 (0) — All Treatment Emergent Adverse Events were reported by treatment regimen and only were not analyzed per intervention.
Rash pustular (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — All Treatment Emergent Adverse Events were reported by treatment regimen and only Treatment Related Treatment Emergent Adverse Events were reported per-intervention since Treatment Emergent Adverse Events were not analysed per intervention.
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) — All Treatment Emergent Adverse Events were reported by treatment regimen and only were not analyzed per intervention.
Headache (Nervous system disorders) | 6 (7) | 5 (6) | 0/0 (0) | 0/0 (0) | 0/0 (0) — All Treatment Emergent Adverse Events were reported by treatment regimen and only were not analyzed per intervention.
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 2 (3) | 0/0 (0) | 0/0 (0) | 0/0 (0) — All Treatment Emergent Adverse Events were reported by treatment regimen and only were not analyzed per intervention.
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0/0 (0) | 0/0 (0) | 0/0 (0) — All Treatment Emergent Adverse Events were reported by treatment regimen and only were not analyzed per intervention.
Toothache (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) — All Treatment Emergent Adverse Events were reported by treatment regimen and only were not analyzed per intervention.
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0) | 0/0 (0) — All Treatment Emergent Adverse Events were reported by treatment regimen and only were not analyzed per intervention.
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0) | 0/0 (0) — All Treatment Emergent Adverse Events were reported by treatment regimen and only were not analyzed per intervention.
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) — All Treatment Emergent Adverse Events were reported by treatment regimen and only were not analyzed per intervention.
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) — All Treatment Emergent Adverse Events were reported by treatment regimen and only were not analyzed per intervention.
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0) | 0/0 (0) — All Treatment Emergent Adverse Events were reported by treatment regimen and only were not analyzed per intervention.
Haematoma (Vascular disorders) | 1 (1) | 2 (4) | 0/0 (0) | 0/0 (0) | 0/0 (0) — All Treatment Emergent Adverse Events were reported by treatment regimen and only were not analyzed per intervention.
Blepharitis (Eye disorders) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0) | 0/0 (0) — All Treatment Emergent Adverse Events were reported by treatment regimen and only were not analyzed per intervention.
Conjunctivitis allergic (Eye disorders) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0) | 0/0 (0) — All Treatment Emergent Adverse Events were reported by treatment regimen and only were not analyzed per intervention.
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0) | 0/0 (0) — All Treatment Emergent Adverse Events were reported by treatment regimen and only were not analyzed per intervention.
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0) | 0/0 (0) — All Treatment Emergent Adverse Events were reported by treatment regimen and only were not analyzed per intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-02-07): https://cdn.clinicaltrials.gov/large-docs/10/NCT03804710/SAP_000.pdf
  • Study Protocol (2018-09-05): https://cdn.clinicaltrials.gov/large-docs/10/NCT03804710/Prot_001.pdf